CLINICAL TRIAL: NCT04164888
Title: A Placebo-controlled, Randomized, Phase 2a, Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of CIVI 007 in Patients on a Background of Stable Statin Therapy
Brief Title: Phase 2a Study to Assess CIVI 007 in Patients on a Background of Statin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Civi Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIVI 007-02-01
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CIVI 007, Dose A (Experimental): Subcutaneous (SC) injection of a PCSK9 inhibitor- low dose given twice
  Interventions: Drug: CIVI 007
- CIVI 007, Dose B (Experimental): SC injection of PCSK9 inhibitor- dose titration
  Interventions: Drug: CIVI 007
- CIVI 007, Dose C (Experimental): SC injection of PCSK9 inhibitor- high dose given twice
  Interventions: Drug: CIVI 007
- Placebo (Placebo Comparator): Placebo SC injection matching PCSK9 inhibitor given twice
  Interventions: Drug: CIVI 007

INTERVENTIONS:
Drug: CIVI 007 — hypercholesterolemia agent

SUMMARY:
Evaluation of the clinical profile (lipid efficacy, safety and PK) across a number of doses of CIVI 007, a PCSK9 inhibitor. Patients to be evaluated will be on a stable background of statin therapy with or without ezetimibe.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index (BMI) between 18.0 and 40.0
2. Stable (>4 weeks prior to the Screening Visit) dose of statin therapy with or without ezetimibe
3. Fasting low-density lipoprotein cholesterol (LDL-C): ≥100 mg/dL for those without cardiovascular disease, or ≥70 mg/dL for those with cardiovascular disease.
4. Fasting triglycerides (TGs) <400 mg/dL

Key Exclusion Criteria:

1. Women who are pregnant, nursing or breast feeding
2. Currently prescribed a lipid lowering agent other than a statin or ezetimibe.
3. Clinically significant disorder or laboratory abnormality that could contraindicate the administration of study drug, affect compliance, interfere with study evaluations, or confound the interpretation of study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Shear, DrPH, Study Director — CiVi Biopharma
Locations (7):
- United States (7):
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Cincinnati, Ohio
  - Research Site, Munroe Falls, Ohio
  - Research Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: CIVI 007, Dose A: Subcutaneous (SC) injection of a PCSK9 inhibitor- low dose given twice
- Experimental: CIVI 007, Dose B: SC injection of PCSK9 inhibitor- dose titration
- Experimental: CIVI 007, Dose C: SC injection of PCSK9 inhibitor- high dose given twice
Period: Overall Study
Arm/Group | Placebo | Experimental: CIVI 007, Dose A | Experimental: CIVI 007, Dose B | Experimental: CIVI 007, Dose C
Started | 12 | 12 | 13 | 12
Completed | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CIVI 007, Dose A | CIVI 007, Dose B | CIVI 007, Dose C | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 12 | 12 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 8 | 8 | 36
  >=65 years | 2 | 3 | 4 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.06) | 56.4 (9.48) | 56.3 (11.63) | 60.3 (8.93) | 57.6 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 6 | 18
  Male | 7 | 9 | 9 | 6 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 13 | 12 | 12 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 3 | 2 | 4 | 12
  White | 9 | 8 | 10 | 8 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Childbearing potential, n [Number; unit: participants] | 1 | 1 | 0 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 171.0 (11.82) | 176.8 (10.58) | 174.9 (9.00) | 170.2 (10.40) | 173.3 (10.54)
Weight [Mean (Standard Deviation); unit: kg] | 89.51 (12.011) | 98.55 (16.473) | 95.30 (18.659) | 82.56 (12.327) | 91.62 (15.924)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 30.75 (4.432) | 31.50 (4.403) | 31.05 (5.306) | 28.56 (3.893) | 30.48 (4.536)
Body mass index category [Count of Participants; unit: Participants]
  less than 30 kg/m2 | 5 | 5 | 5 | 9 | 24
  more or equal to 30 kg/m2 | 7 | 8 | 7 | 3 | 25
PCSK9 [Mean (Standard Deviation); unit: ug/L] | 377.13 (117.819) | 374.03 (106.523) | 467.03 (101.657) | 444.43 (150.172) | 414.81 (123.535)
Fasting LDL-C [Mean (Standard Deviation); unit: mg/dL] | 115.3 (42.49) | 108.2 (27.15) | 102.7 (21.35) | 130.0 (60.39) | 113.9 (40.55)
Taking lower than recommended statin therapy? [Count of Participants; unit: Participants] | 3 | 2 | 2 | 1 | 8
Background statin therapy [Count of Participants; unit: Participants]
  High intensity | 7 | 5 | 7 | 7 | 26
  Moderate intensity | 2 | 6 | 4 | 3 | 15
  Low intensity | 1 | 2 | 0 | 1 | 4
  None | 2 | 0 | 1 | 1 | 4
Ezetimibe use [Count of Participants; unit: Participants] | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Pharmacodynamic Effect of CIVI 007
Description: Percent change from baseline in PCSK9
Time Frame: Baseline, D29, D57, D85
Measure: Median (Full Range); unit: percentage change from baseline
Arm/Group | Placebo | Experimental: CIVI 007, Dose A | Experimental: CIVI 007, Dose B | Experimental: CIVI 007, Dose C
Number analyzed (Participants) | 12 | 12 | 13 | 12
percentage change from baseline
  Day 29 | -4.54 [-15.7 to 63.3] | -71.38 [-89.7 to -63.4] | -76.01 [-92.7 to -18.5] | -82.27 [-93.4 to -48.1]
  Day 57 | -7.42 [-31.6 to 25.8] | -81.08 [-91.0 to -69.9] | -85.48 [-93.0 to -67.6] | -83.42 [-92.2 to -71.2]
  Day 85 | -0.37 [-35.5 to 41.2] | -43.74 [-72.9 to -27.0] | -55.89 [-75.1 to -18.7] | -61.10 [-73.6 to -37.8]
Statistical Analysis 1: Comparison: Placebo vs Experimental: CIVI 007, Dose A; Applying the LOCF method (Last Observation Carried Forward) did not result in any changes at Day 29 or Day 57 due to the lack of missing values and resulted in similar results at Day 85; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -84.56, 95% CI 2-sided [-98.95 to -70.18], Standard Error of Mean 7.137
Statistical Analysis 2: Comparison: Placebo vs Experimental: CIVI 007, Dose B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -80.43, 95% CI 2-sided [-94.58 to -66.29], Standard Error of Mean 7.018
Statistical Analysis 3: Comparison: Placebo vs Experimental: CIVI 007, Dose C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -84.87, 95% CI 2-sided [-99.00 to -70.75], Standard Error of Mean 7.009

2. Secondary Outcome: Assessment of the Lipid Efficacy of CIVI 007
Description: Percent change from baseline in LDL-C
Time Frame: Baseline, Day 29, Day 57, Day 85
Measure: Median (Full Range); unit: percentage change from baseline
Arm/Group | Placebo | Experimental: CIVI 007, Dose A | Experimental: CIVI 007, Dose B | Experimental: CIVI 007, Dose C
Number analyzed (Participants) | 12 | 12 | 13 | 12
percentage change from baseline
  Day 29 | -0.86 [-38.3 to 31.3] | -52.37 [-88.7 to -24.8] | -56.44 [-74.5 to -20.9] | -51.70 [-83.5 to -24.5]
  Day 57 | -10.85 [-57.2 to 42.2] | -51.21 [-71.8 to 27.3] | -61.18 [-82.0 to -14.3] | -59.18 [-82.4 to 1.0]
  Day 85 | -10.08 [-52.4 to 42.2] | -29.66 [-51.9 to 5.7] | -48.65 [-59.1 to 3.3] | -43.51 [-57.1 to 32.7]
Statistical Analysis 1: Comparison: Placebo vs Experimental: CIVI 007, Dose A; Similar changes from baseline were observed for Day 29, Day 57, and Day 85 compared to Day 29, Day 57, and Day 85 LOCF; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -48.03, 95% CI 2-sided [-63.06 to -32.99], Standard Error of Mean 7.460
Statistical Analysis 2: Comparison: Placebo vs Experimental: CIVI 007, Dose B; Similar changes from baseline were observed for Day 29, Day 57, and Day 85 compared to Day 29, Day 57, and Day 85 LOCF; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -49.59, 95% CI 2-sided [-64.50 to 34.69], Standard Error of Mean 7.396
Statistical Analysis 3: Comparison: Placebo vs Experimental: CIVI 007, Dose C; Similar changes from baseline were observed for Day 29, Day 57, and Day 85 compared to Day 29, Day 57, and Day 85 LOCF; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with LOCF; Least Square Mean = -51.99, 95% CI 2-sided [-67.34 to -36.64], Standard Error of Mean 7.616

3. Secondary Outcome: Assessment of CIVI 007 Adverse Events (AEs)
Description: Incidence of any drug-related AEs
Time Frame: Baseline through 2 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Experimental: CIVI 007, Dose A | Experimental: CIVI 007, Dose B | Experimental: CIVI 007, Dose C
Number analyzed (Participants) | 12 | 12 | 13 | 12
Participants
  Mild | 4 | 2 | 5 | 1
  Moderate | 1 | 1 | 3 | 2
  Severe | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 31 weeks.
Arm/Group | CIVI 007, Dose A | CIVI 007, Dose B | CIVI 007, Dose C | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 10/13 | 6/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIVI 007, Dose A (N=12) | CIVI 007, Dose B (N=13) | CIVI 007, Dose C (N=12) | Placebo (N=12)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIVI 007, Dose A (N=12) | CIVI 007, Dose B (N=13) | CIVI 007, Dose C (N=12) | Placebo (N=12)
Alanine aminotransferase increased (Investigations) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 3 (6) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04164888/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04164888/SAP_001.pdf